CLINICAL TRIAL: NCT00070720
Title: Clustered Trial for Improving Perinatal Care in Uruguay/Argentina
Brief Title: Improving Perinatal Care in Latin America
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); Latin American Center for Perinatology (Other); Pan American Health Organization (Other); World Health Organization (Other); Tulane University School of Public Health and Tropical Medicine (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: GN 01; U01HD040477 (NIH)
Record Dates: First submitted 2003-10-07; First posted 2003-10-13 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Episiotomy; Pregnancy
Keywords: Behavior change; Change in practitioner behavior; Episiotomy; Active management of third stage of labor; Global Network; Latin America; Uruguay; Argentina; Maternal and child health; International; Women's health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Opinion Leaders, Academic Detailing, Reminders, and Feedback

SUMMARY:
Many obstetrical interventions used in Latin America, as in other parts of the world, have been shown to be ineffective or harmful, while effective interventions remain underutilized. This study will develop and evaluate an intervention intended to implement two evidence-based practices among birth attendants in Latin America, the selective use of episiotomies and active management of the third stage of labor.

DETAILED DESCRIPTION:
In Latin American countries certain procedures commonly used in obstetrical care (e.g. episiotomy) have been shown to be ineffective or harmful. This study hypothesizes that obstetrical procedures can be changed and new guidelines implemented via peer opinion leader training. It tests an intervention designed to motivate and facilitate health care professionals' development through the implementation and maintenance of simple evidence-based guidelines to increase the use of evidence-based practices by birth attendants at the hospital level in Argentina and Uruguay. The primary outcomes are the use of episiotomies and of oxytocin during the third stage of labor; secondary outcomes include perineal sutures; postpartum hemorrhages; birth attendants' readiness to change status. The sample size was based upon a 10% frequency of oxytocin use and 20% use of episiotomies in the control group. The study hypothesizes a 40% absolute increase in oxytocin use in the intervention group; a 20% absolute reduction in use of episiotomies in the intervention group, calculated at a 0.05 significance level with 80% power.

Following baseline data collections in 24 hospitals, 19 hospitals met inclusion criteria in three urban districts of Argentina and Uruguay and were randomly assigned to an intervention or control group. Baseline data collection has been completed with a total of 6597 single vaginal spontaneous births. The 19 hospitals met inclusion criteria with a rate of active management of third stage of labor under 25% and an episiotomy rate in spontaneous vaginal deliveries above 20%. Opinion leaders in the intervention hospitals have been identified and trained to develop evidence-based guidelines that will be diffused by a multifaceted approach including seminars, academic detailing, reminders, and feedback on utilization rates. The hospitals in the nonintervention group will continue with their standard in-service training activities.

ELIGIBILITY:
Inclusion Criteria for Hospitals

Hospitals were invited to participate in the study if they fulfill the following criteria:

* have an Institutional Review Board (IRB), or existing committee which could serve as such, or have an agreement with an IRB which reviews the research protocols implemented in the hospital;
* have at least 500 vaginal deliveries per year;
* do not have an explicit policy for selective episiotomy and for active management of third stage of labor;
* are located within the study area in Argentina and Uruguay; and
* agree to participate in the study.

Exclusion Criteria for Hospitals

Preselected hospitals are performing baseline data collection. According to the results of the analysis of the baseline data collection, hospitals will be excluded if the episiotomy rate is low or the rate of active management of the third stage of labor is high, according to the following cut-off points:

* Episiotomy rate in spontaneous vaginal deliveries below 20%
* Rate of active management of third stage of labor over 25%

The sample size of the study was increased to allow for exclusions.

Expectant management is defined as "a hands-free policy" during third stage of labor until the placenta is expelled: no use of uterotonics or special maneuvers.

Sampling, Recruitment, and Screening Procedures

Latin American Center for Perinatology (CLAP) coordination team will be responsible for the hospital selection. The hospitals' fulfillment of selection criteria will be obtained through a survey of the Heads of the Obstetrical Departments.

Besides the selection criteria, the coordination unit will invite the hospitals to participate according to:

* their participation in previous trials coordinated by CLAP,
* their participation in other trials or research activities, and
* their location.

Of particular interest are the characteristics of each preselected hospital regarding the structure of the professional staff, number of deliveries, and clinical guidelines policy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21780
Dates: Start 2003-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Episiotomies
Oxytocin use in third stage of labor

SECONDARY OUTCOMES:
Perineal sutures
Postpartum hemorrhage
Birth attendants' readiness to change status

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Buekens, MD, PhD, Principal Investigator — Tulane School of Public Health and Tropical Medicine
Locations (1):
- Hospital de Clinicas, Montevideo, Uruguay

REFERENCES:
- [Background] Althabe F, Buekens P, Bergel E, Belizan JM, Kropp N, Wright L, Goco N, Moss N; for the Guidelines Trial Group. A cluster randomized controlled trial of a behavioral intervention to facilitate the development and implementation of clinical practice guidelines in Latin American maternity hospitals: the Guidelines Trial: Study protocol [ISRCTN82417627]. BMC Womens Health. 2005 Apr 11;5(1):4. doi: 10.1186/1472-6874-5-4. PMID 15823211
- [Background] Kropp N, Hartwell T, Althabe F. Episiotomy rates from eleven developing countries. Int J Gynaecol Obstet. 2005 Nov;91(2):157-9. doi: 10.1016/j.ijgo.2005.07.013. Epub 2005 Oct 5. No abstract available. PMID 16169552
- [Derived] Althabe F, Buekens P, Bergel E, Belizan JM, Campbell MK, Moss N, Hartwell T, Wright LL; Guidelines Trial Group. A behavioral intervention to improve obstetrical care. N Engl J Med. 2008 May 1;358(18):1929-40. doi: 10.1056/NEJMsa071456. PMID 18450604
- See also: Tulane School of Public Health and Tropical Medicine — http://www.sph.tulane.edu/
- See also: RTI International — http://www.rti.org/
- See also: Institute for Clinical Effectiveness and Health Policy (IECS) — http://www.iecs.org.ar